CLINICAL TRIAL: NCT06444893
Title: Morphofunctional Analysis, Gene Expression of Inflammation Molecules and Response Mechanisms to Oxidative Stress in Kidney Tissue of Deceased Patients With COVID-19: "Ancestral Variant"
Brief Title: Morphofunctional, Gene, Inflammation Molecules and Oxidative Stress Analysis in Kidney Tissue of COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Jesus Rivero, MD, Principal Investigator, Instituto Nacional de Enfermedades Respiratorias
Other Study IDs: C-5920
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Kidney Injury; Gene Amplification; Oxidative Stress; Inflammatory Response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — kidney biopsies of deceased patients with COVID-19
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The involvement of the kidneys in patients infected with the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at the outset of the pandemic was associated with high mortality rates worldwide. This was in part due to the generation of an inflammatory process and exacerbated oxidative stress. The present study was initiated to investigate the relationship between morphofunctional changes and gene expression in the kidney tissue of deceased Mexican patients prior to the initiation of vaccination.

The investigator designed a single-center, prospective, cohort study, to analyze and relate the morphofunctional changes and gene expression of inflammatory and oxidative stress molecules in the kidney tissue of men who died from severe COVID-19. A total of 40 percutaneous renal biopsies from deceased patients with severe acute respiratory syndrome coronavirus 2 infection were included in the study and divided into two a groups. One group was preserved in trizol to obtain RNA and total protein, while the remaining sample was fixed in formalin to be examined by staining with hematoxylin and eosin. The histopathological analysis was conducted by an experienced pathologist. The expression of molecules was evaluated by real-time polymerase chain reaction assay (nphs2, slc9a1, cx3cl1, havcr1, slc22a17, sod2, egf, timp2, hmox1, fabp1, and so forth). The following biomarkers were analyzed: interleukin-6, Arginase-1 (Arg-1), Dipeptidyl peptidase-4 (DPP-4), GSTT1, type I gamma-glutamyltransferase (GGT1), Occludin (OCL), CYP3A4, and Claudin-8 (CL-8). Additionally, Western blot analysis was conducted on claudin-5 (CL-5), occludin, HSP70, Nuclear factor erythroid 2-related factor-2 (NRF-2), superoxide dismutase-2 (SOD-2), nicotinamide adenine dinucleotide phosphate dehydrogenase 1 (NQO1), Gamma glutamylcysteine synthase (γ-GCL), and receptor for advanced glycation end products (RAGE). The estimated glomerular filtration rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, with the subjects divided into two groups based on their eGFR: >60 or <60 ml/min/1.73 m². The statistical analysis was conducted using the Stata program and GraphPad software, version 10.2.3.

ELIGIBILITY:
Inclusion Criteria:

* Not having at least one creatinine measurement.
* Family members will not accept to participate.

Exclusion Criteria:

* Specimens with sub-optimal quality for analysis.

Ages: 15 Years to 80 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The investigators chose only males for the study due to they presented a major deleterious effect in scientific literature.
Study Population: Adults >15 years old who died at the INER with a confirmed diagnosis of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
Fibrosis and sclerosis scores for identifying morphological changes in kidney tissue. | From the date of postmortem kidney biopsy until the date of histopathological report, in average seven days.
  Morphological changes were evaluated by the fibrosis and sclerosis scores (mild, moderate and severe), using direct visualization of nephron compartments (glomerular and tubulointerstitial) of patients who died due to severe COVID-19.
The estimated glomerular filtration rate for evaluating functional changes. The estimated glomerular filtration rate for evaluating functional changes. | From the date of arrival at the hospital until the date of death, in average one month.
  Functional changes were calculated using the estimated glomerular filtration rate (> 60 vs < 60 ml/min/1.73m2) of patients who died due to severe COVID-19.

SECONDARY OUTCOMES:
Differential gene expression using polymerase chain reaction | From the date of postmortem kidney biopsy until the date of measure of differential gene expression, evaluated in 72 months.
  Changes in differential gene expression in the kidney tissue of patients who died from due to severe COVID-19.
Quantity of inflammatory molecules expressed in picograms of proteins. | From the date of postmortem kidney biopsy until the date of measure the inflammatory molecules expressed in the tissue, evaluated in 72 months.
  Changes in the quantity of inflammatory molecules in the kidney tissue of patients who died due to severe COVID-19.
Quantity of oxidative stress molecules expressed in picograms of proteins. | From the date of postmortem kidney biopsy to the date of measure of oxidative stress molecules expressed in the tissue report, evaluated in 72 months.
  Changes in the quantity of oxidative stress molecules expressed in the kidney tissues of patients who died due to severe COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Respiratory Diseases, Mexico City, Mexico City, Mexico